CLINICAL TRIAL: NCT02348047
Title: Randomized Study Comparing the ASV to Conventional Ventilation for Intubated Patients During Inter-hospital Transfers. Controlled Randomized Monocentric Prospective Study Comparing ASV Versus Conventional Ventilation Modes
Brief Title: (S5-SAMU) Randomized Study Comparing the ASV (Adaptative Support Ventilation) to Conventional Ventilation
Acronym: S5-SAMU
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: PI resignation
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Collaborators: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-CH-01
Record Dates: First submitted 2015-01-16; First posted 2015-01-28 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional ventilation (Active Comparator): Conventional ventilation - manual mode
  Interventions: Device: Hamilton T1
- ASV (Experimental): Intellivent ASV ( Adaptative Support Ventilation )Ventilation- automatic mode
  Interventions: Device: Hamilton T1

INTERVENTIONS:
Device: Hamilton T1

SUMMARY:
Compare ventilation parameters in Adaptative Support Ventilation mode to conventional mode, on intubated, ventilated and sedated patients, during their secondary transfer from an hospital to another, by a SMUR team.

ELIGIBILITY:
Inclusion Criteria:

* Intubation
* Secondary transfer (interhospital)
* Informed patients / close relations, signed consent

Exclusion Criteria:

* Primary transport of a ventilated, intubated, sedated patient
* Patient in limitation and stop of active therapeutics, dying person
* Broncho pleural fistula
* Patient under ECMO
* Patient included in another research submitted to consent
* Supervision, loss of liberty
* Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-03-11 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Ventilation parameter: VT | Participants are followed during their inter hospital transfer,an expected average of 1 or 2 hours"
Ventilation parameter: respiratory rate | Participants are followed during their inter hospital transfer,an expected average of 1 or 2 hours"
Ventilation parameters: Fi02 | Participants are followed during their inter hospital transfer,an expected average of 1 or 2 hours"
Ventilation parameter: PEEP | Participants are followed during their inter hospital transfer,an expected average of 1 or 2 hours"
Ventilation parameter: ETC02 | Participants are followed during their inter hospital transfer,an expected average of 1 or 2 hours"

SECONDARY OUTCOMES:
Numbers of manual adjustments | Participants are followed during their inter hospital transfer,an expected average of 1 or 2 hours"

CONTACTS AND LOCATIONS:
Overall Officials: Marilyne ROTI BOUNY, MD, Principal Investigator — Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer
Locations (1):
- Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer, Service d'infectiologie, Toulon, France